CLINICAL TRIAL: NCT00390572
Title: Sleep Specialty Consultation: Improving Management of Sleep Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 05-213; 0016 (Other Grant/Funding Number: VA R&D); 01147 (Other Grant/Funding Number: VA R&D)
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Disorders
Keywords: sleep; consultation and referral; outcome assessment; primary care
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Specialty Consultation (Experimental): Participants randomized to receive a one-time sleep consultation at beginning of study
  Interventions: Behavioral: Sleep Specialty Consultation
- Treatment as Usual (No Intervention): Participants randomized to receive a one-time sleep consultation after completing study procedures (after 10 month study wait-list period).

INTERVENTIONS:
Behavioral: Sleep Specialty Consultation — The Sleep Specialty Consultation (SSC) consisted of: (1) a thorough sleep disorders evaluation accomplished via a clinician-administered structured interview designed to assess specific symptoms of global sleep disorder categories, review of a sleep history questionnaire, and review of available (CPRS) medical/psychiatric electronic records; (2) education about the specific sleep disorders diagnoses and relevant treatment recommendations provided to the patients; and (3) standardized diagnostic information and treatment recommendations provided to the participants' primary care providers.
  Arms: Sleep Specialty Consultation

SUMMARY:
Sleep disorders are prevalent health problems that reduce quality of life, increase risks for medical disease, and enhance healthcare costs/utilization. Only a small proportion of these cases are diagnosed in primary care. Pilot data from this VA suggest that sleep disorders are not adequately managed in a primary care setting: 33% of veterans with an insomnia complaint had an undiagnosed primary sleep disorder (e.g., sleep apnea), and 50% of these patients were prescribed pharmacologic treatment for insomnia by their primary care providers.

DETAILED DESCRIPTION:
Sleep disorders are prevalent health problems that reduce quality of life, increase risks for medical disease, and enhance healthcare costs/utilization. Only a small proportion of these cases are diagnosed in primary care. Pilot data from this VA suggest that sleep disorders are not adequately managed in a primary care setting: 33% of veterans with an insomnia complaint had an undiagnosed primary sleep disorder (e.g., sleep apnea), and 50% of these patients were prescribed pharmacologic treatment for insomnia by their primary care providers. This project tests the incremental benefits of adding a one-time sleep specialty consultation (SSC) to usual primary care for reducing sleep disturbance, diurnal dysfunction, quality of life concerns and health care utilization among veterans enrolled in the DVAMC Primary Care Clinics. The SSC will consist of: (1) a thorough sleep disorders evaluation accomplished via a clinician-administered structured interview designed to assess specific symptoms of global sleep disorder categories, review of a sleep history questionnaire, and review of available (CPRS) medical/psychiatric electronic records; (2) education about the specific sleep disorders diagnoses and relevant treatment recommendations provided to the patients; and (3) standardized diagnostic information and treatment recommendations provided to the participants' primary care providers. Study hypotheses predict that patients who receive an SSC with feedback to their primary care providers will show greater improvements in sleep, mood, quality of life, and patient satisfaction, as well as larger reductions in health care utilization than will those who receive usual care alone. This is a randomized, wait-list control, clinical intervention study of 300 veterans with sleep complaints. Eligibility criteria include: sleep complaint for > 1 month duration, Pittsburgh Sleep Quality Index score > 5; mental status score > 24 on Folstein MMSE, no unstable medical or psychiatric disorder, and approval of primary provider. The SSC intervention consists of a clinician-administered structured interview assessing sleep pathology, plus manualized feedback to patients and primary care providers. Participants are randomly assigned to SSC or Wait List Control (WLC) conditions. Measures of sleep, mood, quality of life, and patient satisfaction are obtained at enrollment and at 5- and 10-month follow-up. Computerized utilization data is obtained for the 10 months prior to and 10 months following enrollment. A series of multivariate and univariate statistical tests will be conducted.

Study findings should provide important new information about managing both the sleep problems and overall health care utilization patterns of patients with sleep complaints presenting in VA primary care settings. If SSC-evaluated patients show substantial reductions in their VA inpatient/outpatient utilization, this finding could have important cost-saving implications to the VA system.

ELIGIBILITY:
Inclusion Criteria:

* veteran seen at Durham VAMC for primary care;
* must have had a sleep complaint for > 1 month;
* not being treated by a sleep specialist for sleep complaint;
* provide informed consent;
* have concurrence for enrollment from their assigned MD PCP;
* score >5 on the Pittsburgh Sleep Quality Index at time of screening

Exclusion Criteria:

* terminal illness;
* acute or highly unstable Axis I psychiatric condition;
* not mentally competent;
* unstable living environment;
* unstable medical or psychiatric condition;
* established sleep disorder or currently under the care of one or more of our VAMC's sleep disorders specialists;
* previous evaluation by sleep disorders specialist;
* refuse to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-01; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Olsen MK, Stechuchak KM, Edinger JD, Ulmer CS, Woolson RF. Move over LOCF: principled methods for handling missing data in sleep disorder trials. Sleep Med. 2012 Feb;13(2):123-32. doi: 10.1016/j.sleep.2011.09.007. Epub 2011 Dec 14. PMID 22172964
- [Result] Edinger JD, Ulmer CS, Grubber J, Zervakis JB, Olsen MK. Effects of a One-Time Sleep Specialty Consultation on Sleep Problem Management in Primary Care. [Abstract]. Sleep. 2011 Oct 20; 34(Suppl):A337,0984.
- [Result] Zervakis JB, Ulmer CS, Edinger JD. Can a One-Time Sleep Specialty Consultation Enhance Providers' Attention to Sleep Problems in Primary Care? [Abstract]. Sleep. 2010 Mar 1; 33(Suppl):A365,1092.
- [Derived] Edinger JD, Grubber J, Ulmer C, Zervakis J, Olsen M. A Collaborative Paradigm for Improving Management of Sleep Disorders in Primary Care: A Randomized Clinical Trial. Sleep. 2016 Jan 1;39(1):237-47. doi: 10.5665/sleep.5356. PMID 26285003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 156 subjects were consented and enrolled in the study, but 15 were excluded before randomization for not meeting entry criteria and 4 withdrew because they found study procedures too demanding. The remaining 137 continued in the study and were randomly assigned.
Period: Overall Study
Arm/Group | Sleep Specialty Consultation | Treatment as Usual
Started | 68 | 69
Completed | 60 | 64
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 8 | 4
Not completed — health condition | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat: All participants who were randomized to treatment condition.
Groups:
- Sleep Specialty Consultation: Participants randomized to receive a one-time sleep consultation at beginning of study
  Sleep Specialty Consultation: The Sleep Specialty Consultation (SSC) consisted of: (1) a thorough sleep disorders evaluation accomplished via a clinician-administered structured interview designed to assess specific symptoms of global sleep disorder categories, review of a sleep history questionnaire, and review of available (CPRS) medical/psychiatric electronic records; (2) education about the specific sleep disorders diagnoses and relevant treatment recommendations provided to the patients; and (3) standardized diagnostic information and treatment recommendations provided to the participants� primary care providers.
- Total: Total of all reporting groups
Arm/Group | Sleep Specialty Consultation | Treatment as Usual | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (13.7) | 55.9 (13.4) | 55.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 54 | 54 | 108
Region of Enrollment [Number; unit: participants]
  United States | 68 | 69 | 137

OUTCOME MEASURES:

1. Primary Outcome: Provider Adherence to Sleep Specialist Recommendations
Description: Provider outcomes included the provider's number of participant sleep lab referrals, referrals to other specialty clinics for evaluation/treatment participant sleep problems, and presence of newly initiated sleep-focused therapies for participants. Information about these outcomes was obtained via review of provider orders and information included in notes entered into the VA's computerized medical record system (CPRS). To quantify this outcome, the number of participants referred by providers for sleep-focused diagnostic tests and interventions was compared across arms.
Time Frame: 10 months after baseline
Population: Data was included for all participants.
Measure: Number; unit: participants
Arm/Group | Sleep Specialty Consultation | Treatment as Usual
Number analyzed (Participants) | 68 | 69
participants
  Ferritin Level Check Ordered | 4 | 0
  Sleep Clinic Referral | 8 | 4
  Polysomnography Referral for Apnea | 32 | 3
  Polysomnography Referral for Any Reason | 33 | 4
  Mental Health Clinic Referral | 13 | 4
  Posttraumatic Stress Disorder Clinic Referral | 1 | 1
  Substance Abuse Outpatient Clinic Referral | 4 | 1

2. Primary Outcome: Diary Sleep: Total Wake Time and Total Sleep Time
Description: Changes in sleep from baseline to subsequent follow-up periods were evaluated using both actigraphy and electronic diaries via a personal digital assistant (PDA). Primary outcome measures derived from the PDA included total sleep time (TST), total wake time (TWT: SOL+WASO), and sleep efficiency (SE). Wrist Actigraphy. Mini-Mitter® Actiwatch actigraphs were used to derive the primary objective estimates of TST, TWT, and SE. Mean values of TST, TWT and SE were obtained for each participant at baseline, 5 months and 10 months post-randomization and served as the actigraphic dependent measures in study analyses.
Time Frame: 10 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sleep Specialty Consultation | Treatment as Usual
Number analyzed (Participants) | 68 | 69
minutes
  Total Sleep Time | 401.2 (69.9) | 397.0 (75.9)
  Total Wake Time | 59.7 (42.0) | 79.6 (58.7)

3. Secondary Outcome: Sleepiness
Description: Changes in subjectively assessed daytime sleep propensity were measured using the Epworth Sleepiness Scale (ESS), a commonly employed in both sleep research and clinical applications. The ESS items inquire about the chance of dozing off in each 8 different situations. Responses are rated on a 4 point scale reflecting the respondents perceived likelihood of falling asleep. To quanitfy this outcome, the percentage of participants achieving normal sleep (less than 10 on ESS) was compared across arms at 10 months.
Time Frame: 10 months
Measure: Number; unit: percentage of participants
Arm/Group | Sleep Specialty Consultation | Treatment as Usual
Number analyzed (Participants) | 68 | 69
percentage of participants | 69 | 50

4. Primary Outcome: Sleep Efficiency
Description: as for outcome 2
Time Frame: 10 Months after Baseline
Population: Data from all participants was included.
Measure: Mean (Standard Deviation); unit: percentage of time in bed spent sleeping
Arm/Group | Sleep Specialty Consultation | Treatment as Usual
Number analyzed (Participants) | 68 | 69
percentage of time in bed spent sleeping | 87 (9.7) | 83.5 (11.7)

5. Primary Outcome: Sleep Quality
Description: Changes in overall sleep quality were evaluated using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-rating scale that yields a quantitative index of general sleep quality/disturbances. The PSQI is composed of 4 open-ended questions and 19 self-rated items (0-3 scale) assessing sleep quality and disturbances over a 1-month interval. The PSQI yields a global score of sleep quality ranging from 0 to 21. A score of <= 5 on the PSQI is considered normal sleep quality.
Time Frame: 10 Months
Population: Data from all participants were included in analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sleep Specialty Consultation | Treatment as Usual
Number analyzed (Participants) | 68 | 69
units on a scale | 8.3 (3.7) | 9.5 (3.5)

ADVERSE EVENTS:
Arm/Group | Sleep Specialty Consultation | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69
Other Adverse Events (participants affected / at risk) | 0/68 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No